CLINICAL TRIAL: NCT02118389
Title: The Effect of Meal Replacement Beverage(Glucerna) on Body Composition,Lipid Metabolism and Blood Pressure in Patients With Obesity
Brief Title: Effect of Meal Replacement Beverage(Glucerna) on Body Composition,Lipid Metabolism and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Professor, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Glucerna
Record Dates: First submitted 2014-04-01; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2013-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucerna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glucerna,Meal Replacement (Experimental): Glucerna 52g instead of night meal 5weeks
  Interventions: Dietary Supplement: Glucerna

INTERVENTIONS:
Dietary Supplement: Glucerna — Glucerna 52g meal replacement
  Other Names: Glucerna （Abbort，SR）

SUMMARY:
Effect of Meal Replacement Beverage(Glucerna) on Body Composition,lipid metabolism and blood pressure

DETAILED DESCRIPTION:
The Effect of Meal Replacement Beverage(Glucerna) on Body Composition,lipid metabolism and blood pressure in Patients with Obesity

ELIGIBILITY:
Inclusion Criteria:

1. age：14~60years
2. BMI ≥ 28kg/m2
3. without liver, kidney, gastrointestinal and other major organic serious diseases,lactating women, pregnancy

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Dual energy X-ray absorptiometry | 5 weeks

SECONDARY OUTCOMES:
lab testing | 5weeks

OTHER OUTCOMES:
blood pressure | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qu Shen, PhD, Study Director — Shang Tenth People's Hospital